CLINICAL TRIAL: NCT02483013
Title: Clinical, Controlled, Double-blind Study on the Effect of Whitening Dentifrices on Tooth Color and Tooth Sensitivity
Brief Title: Clinical Study of the Whitening Dentifrices on Tooth Color and Sensitivity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Camila Tirapelli, PhD, University of Sao Paulo
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 01546412.4.0000.5419
Record Dates: First submitted 2015-06-15; First posted 2015-06-26 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Dentin Hypersensitivity
Keywords: whitening dentifrices; color alteration; tooth sensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — sorriso

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Whitening dentifrices (Active Comparator): Two groups used whitening dentifrices, three times per day during four weeks
  Interventions: Other: whitening dentifrices
- Placebo (Placebo Comparator): One group used conventional dentifrice, three times per day during four weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Other: whitening dentifrices — Two groups: participants received the instructions to use only the blinded supplied whitening dentifrice (Colgate Luminous White® or Close up White Now®) and toothbrush to make the habitual oral hygiene, three times per day during four weeks
  Other Names: Colgate Luminous White®; Close up White Now®
  Arms: Whitening dentifrices
Other: Placebo — One group: participants received the instructions to use only the blinded supplied non-whitening dentifrice (Sorriso®) and toothbrush to make the habitual oral hygiene, three times per day during four weeks
  Other Names: Sorriso®
  Arms: Placebo

SUMMARY:
Objective:The aim of this clinical study was to evaluate tooth color alteration (ΔE) and tooth sensitivity (TS) in patients that used two commercial brand-whitening dentifrices for four weeks. Sixty participants were selected in accordance with inclusion and exclusion criteria and randomly allocated in three groups (n=20): G1-Colgate Luminous White®, G2- Close up White Now® and G3- Sorriso® dentifrice (placebo). Then, participants received the instructions to use only the blinded supplied dentifrice and toothbrush to make the habitual oral hygiene, three times per day during four weeks. Evaluators assessed tooth color (CIEL*a*b system) and TS (VAS scale) at baseline and every week (assessment points 1, 2, 3 and 4). Two-way ANOVA and posterior Tukey and Friedman test analyzed data (α = 0.05).

ELIGIBILITY:
Inclusion Criteria:

* At least six anterior teeth without restorations
* Participants should have good general and oral health (no dental caries and periodontal disease)

Exclusion Criteria:

* Tooth sensitivity
* Any condition that could cause tooth sensitivity (non-carious cervical lesions, dentin exposure)
* Participants following orthodontic treatment
* Smokers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-08; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Tooth color | 4 weeks
  Tooth color was measured by Vita Easyshade spectrophotometer over a 4 weeks time frame.
Tooth sensitivity | 4 weeks
  The pain caused by dentin hypersensitivity was measured over a 4 weeks time frame. The investigators stimulated the cervical region of the teeth with a blast of air from a triple syringe and patients reported pain intensity in accordance to Visual Analogue Scale (0= no pain, 10= pain bad as can be).

CONTACTS AND LOCATIONS:
Overall Officials: Camila Tirapeli, PhD, Principal Investigator — University of Sao Paulo Ribeirão Preto Campus
Locations (1):
- University of Sao Paulo, Ribeirao Preto Campus, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- See also: Dental School of Ribeirão Preto website — http://www.forp.usp.br